CLINICAL TRIAL: NCT03002168
Title: A Single Center, Randomized, Double-blind, Placebo Controlled, Two-way Crossover Study to Determine the Fat Losses in Stool Associated With Alpha-CD Use as Compared to Placebo Using a Radiotracer
Brief Title: Determining Lipid Content in Stool After Alpha-cyclodextrin
Acronym: FMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: SFI Research (Industry)
Responsible Party: Principal Investigator, Michael D. Jensen, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-005006
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Healthy Participants
MeSH Terms: interventions — alpha-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-cyclodextrin (Active Comparator): Two 1 gram Alpha-cyclodextrin tablets given per fat-containing meal. A total of 6 tablets (6 grams) per day for the first two consecutive days of active treatment period. Triolein radiolabeled with 100 microcuries of 3^Hydrogen and Tripalmitin radiolabeled with 20 microcuries of 14^Carbon given orally with liquid breakfast meal.
  Interventions: Dietary Supplement: Alpha-cyclodextrin; Radiation: Triolein radiolabeled with 100 microcuries of 3^Hydrogen; Radiation: Tripalmitin radiolabeled with 20 microcuries of 14^Carbon
- Placebo (Placebo Comparator): Two Placebo Alpha-cyclodextrin tablets given per fat-containing meal. A total of 6 tablets per day for the first two consecutive days of placebo treatment period.Triolein radiolabeled with 100 microcuries of 3^Hydrogen and Tripalmitin radiolabeled with 20 microcuries of 14^Carbon given orally with liquid breakfast meal.
  Interventions: Dietary Supplement: Placebo; Radiation: Triolein radiolabeled with 100 microcuries of 3^Hydrogen; Radiation: Tripalmitin radiolabeled with 20 microcuries of 14^Carbon

INTERVENTIONS:
Dietary Supplement: Alpha-cyclodextrin — Alpha-cyclodextrin is approved by the Food and Drug Administration as a dietary ingredient.
  Other Names: FBCx; Calorease
  Arms: Alpha-cyclodextrin
Dietary Supplement: Placebo — Placebo tablets identical in appearance to the active comparator
  Arms: Placebo
Radiation: Triolein radiolabeled with 100 microcuries of 3^Hydrogen — A MicroCurie (µCi) is a measure of radioactivity.
Radiation: Tripalmitin radiolabeled with 20 microcuries of 14^Carbon — A MicroCurie (µCi) is a measure of radioactivity.

SUMMARY:
The Investigator hypothesizes that the currently used dose of dietary ingredient alpha-cyclodextrin (α-CD) will result in greater loss of dietary fat in the stool compared with placebo. The proposed studies will address the degree to which α-CD increases dietary fat loss.

The Investigator will conduct the study and analyze the samples at Mayo Clinic in Rochester, Minnesota.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo controlled, two-way crossover trial in healthy volunteers. The primary objective is to determine the fat losses in stool associated with alpha-cyclodextrin use as compared to placebo using a radiotracer. The study design will include two treatment periods, assigned in random order:

* Treatment 1 consists of subjects receiving α-CD and a meal containing the fatty acid radiotracers
* Treatment 2 consists of subjects receiving placebo and a meal containing the fatty acid radiotracers

All subjects randomized to receive α-CD will orally ingest two tablets containing α-CD, or placebo, with a standardized liquid breakfast (100 µ Ci of [3H]triolein and 20 µ Ci of [14C] tripalmitin). The tablets will be consumed with 150 ml of still (uncarbonated) water immediately prior to consuming each meal.

Subjects will be observed for a period of 48 hours as an in-patient, and then an additional 24 hours as an out-patient following the breakfast meal containing the radiotracers. During this time the participants will undergo a meal fatty acid metabolism study, through hourly blood and fecal sampling, to assess meal fatty acid oxidation and storage.

The participants will then undergo a further ≥ 14 day washout period before crossing over to the alternate treatment, where all evaluations will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy weight stable individuals (defined as a Body Mass Index (BMI) of ≥18.5 and <27, and stable for at least the preceding two months from Screening).
* Not pregnant, and if of childbearing potential, agrees to use adequate birth control (hormonal or barrier method of birth control or abstinence) prior to study entry and during the trial and agrees not to donate sperm or ova, for the duration of the study
* Subjects ≥18 and ≤60 years of age at screening
* Consistent regular bowel movement (defined as between 3 times a day, to 1 time per day)
* Provide Informed Consent
* Willing and able to complete study procedures within the study timelines
* Adequate renal function: serum creatinine less than 1.5 x Upper Limit of Normal (ULN)
* Adequate liver function: serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) and serum glutamic pyruvic transaminase/alanine aminotransferase (SGPT/ALT) ≤ 2 × ULN and serum bilirubin ≤ 1.5 × ULN, unless Gilbert's syndrome has previously been confirmed for the subject
* Adequate bone marrow function: white blood cells (WBCs) ≥ 3,000/mm^3, absolute neutrophil count (ANC) ≥ 1,500/mm^3, hemoglobin ≥ 9 gram/deciLiter, and platelets ≥ 100,000/mm^3

Exclusion Criteria:

* Evidence of chronic pancreatitis
* Evidence of irritable bowel syndrome (medical or self-diagnosed)
* Previous gallbladder surgery
* Use of enemas and/or suppositories within 30 days of Screening
* Consuming ≥ 375 mg of caffeine per day (equivalent to 5 serves of 1 oz. restaurant style espresso per day)
* History of febrile illness within 5 days prior to Screening
* Evidence or history of substance or alcohol abuse
* History of major depression, bipolar disorder, or schizophrenia (per DSM4 criteria; Diagnostic and Statistical Manual of Mental Disorders)
* Current use of prescription or non-prescription weight loss products (≥ 2 week washout period is required to become eligible)
* Smoking ≥ 20 cigarettes (~one pack) per week
* Significant dietary restrictions (incl. vegan, vegetarian diets and any subject not prepared to consume any of the standardized food/s)
* Evidence of an active eating disorder (incl. anorexia nervosa, bulimia, and/or obsessive compulsive disorders)
* Use of other investigational agent(s at the time of enrollment, or within 30 days or five half-lives of enrollment, whichever is longer
* Pregnant or lactating
* Current use of any medication known to affect gut motility
* History of malignancy, treated or untreated, within the past five years, with the exception of non-melanoma skin cancer and cervical carcinoma in situ
* A known history of hypersensitivity to any of the α-CD ingredients
* Any other health condition that would preclude participation in the study in the judgment of the principal investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Change in lipid content in stool, measured using 3^H radiolabeled tracer | Baseline, 6 hours

SECONDARY OUTCOMES:
Change in lipid content in stool, measured using 14^C radiolabeled tracer | Baseline, 6 hours
Change in blood triglyceride concentrations, measured using 3^H radiolabeled tracer | Baseline, 6 hours
Change in blood triglyceride concentrations, measured using 14^C radiolabeled tracer | Baseline, 6 hours
Change in blood glucose concentration | Baseline, 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lytle KA, Harteneck DA, Noble AM, Jensen MD. The Soluble Fiber alpha-Cyclodextrin Does Not Increase the Fecal Losses of Dietary Fat in Adults-A Double-Blind, Randomized, Placebo-Controlled, Crossover Trial. J Nutr. 2018 Sep 1;148(9):1421-1425. doi: 10.1093/jn/nxy135. PMID 30107536